CLINICAL TRIAL: NCT04293367
Title: Fuel Utilization, Diet Composition, and Exercise in African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jeanine Albu, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLR 1-10-CT-01; #: 1-10-CT-01 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Diabetes; Insulin Resistance
Keywords: Obesity; Prediabetes; metabolic flexibility; insulin sensitivity; high-intensity interval training; exercise tolerance
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance; Prediabetic State | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The study team will conduct a randomized clinical trial in 48 healthy pre-menopausal sedentary overweight and obese African American women. The women will be randomized to two groups: a) half of the women in each diet group will be training (EX) and b) half of the women in each diet group will be sedentary (C). Each woman will participate over a 5 months period, through 4 menstrual cycles so that baseline and post-intervention measurements are done during the follicular phase of the menstrual cycle. The baseline and post-intervention measurements will be done after a 10-day period of controlled eucaloric High-Fat feeding. On Days 9-11 of the 10 -day period they will be in-patients in the CRR and they will all be sedentary. On Day 9 they will be admitted to the Metabolic Chamber and have 24-hour energy expenditure measurements as previously described which will be used for the diet on subsequent days in the CRR. On Day 10 they will be fed the same amount of calories they bu
Who Masked: Participant, Investigator
Masking Description: Potential subjects will be from an African American descent which will be defined as having all four grandparents reported as African Americans. The subjects will be healthy (blood work, Hx and PE), non-diabetic (OGTT) pre-menopausal, age range 20-40 years, BMI range of 25-40, with regular menstrual periods, sedentary (exercise no more than 2 times/week, for one hour or spend no more than 1000 - 1500 Kcal/wk in physical activity as determined by a Paffenbarger questionnaire). Subjects will be excluded if there is any indication what so ever that they have any cardiac or pulmonary illnesses which may interfere with their capacity to exercise, if they are smokers, consume more than 2 oz. of ethanol/day, have had a weight change greater than + 2 kg in the past 3 months, are currently taking medications or have any physical conditions which may affect insulin action and/or lipid metabolism or have hyperlipidemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 14 African American Women with obesity will be randomly assigned to the 14-week high intensity interval training program
  Interventions: Other: High Intensity Interval Training (HIIT)
- Control (No Intervention): 14 African American Women with obesity will be randomly assigned to serve as a reference group, i.e. follow the same protocol as the experimental group, however, they will not undergo exercise training

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — HIIT involves exercising in blocks of time (typically 4-5 minutes) where a small percentage of the time (typically 1 minute) is spent above the anaerobic (lactate) threshold (the "work interval") followed by the remainder of the time at a sub-anaerobic threshold ("active recovery").
  Arms: Exercise

SUMMARY:
African American women have a high prevalence of obesity and type 2 diabetes and do not optimally burn fat and carbohydrates in response to changes in these nutrients in their diets. This research project seek to determine if high intensity interval training (HIIT) exercise training can help healthy, but inactive, premenopausal, non-diabetic women increase their bodies' use of fat and carbohydrates when provided with a high fat or low fat diets. In this study, investigators will measure the rate at which fat is burned in response to weight maintaining low-fat and high-fat diets and how exercise may affect these responses.

DETAILED DESCRIPTION:
African Americans have the highest age-adjusted death rate for heart disease and diabetes in the United States. Obesity, a significant risk factor for these conditions, is highly prevalent in African Americans, particularly women, leading to increased co-morbidities. Cardiovascular risk and incidence were reported to be higher in African American women than in both white women and African American men. Ethnic differences in lifestyle behaviors and economic disadvantage account for some of this disparity but genetic/molecular factors may play a role. The study team has shown that more pre-menopausal, non-diabetic, African American women do not increase post-absorptive lipid oxidation in response to a eucaloric increase in dietary fat than white women counterparts. African American women were also shown to have increased rates of low aerobic capacity (VO2peak) and insulin resistance.

A lack of increasing fuel utilization in response to an increase in fuel availability, particularly fat, is associated with obesity and insulin resistance and is attributed to a decrease in the oxidative capacity of the skeletal muscle. An eucaloric increase in dietary fat leads to increased post-absorptive lipid utilization through hormonal changes that affect the mitochondria and a decrease in this response is postulated to reflect a decrease in the mitochondria/oxidative capacity. Lipid utilization in response to an increase in dietary fat is enhanced by acute exercise. Aerobic training could also improve aerobic capacity and insulin resistance and increases the oxidative capacity/mitochondrial activity in the skeletal muscle, measured in vitro. The degree to which training affects aerobic capacity and metabolism differs with the type, intensity and duration of training and with the population studied. High-intensity interval training (HIIT) programs improved aerobic fitness and insulin resistance in cardiac, sedentary and obese individuals and rapidly increased markers of lipid oxidation and mitochondrial activity in skeletal muscle, measured in vitro. A great appeal of HIIT is that lesser time per week spent exercising may be needed to produce these effects. There have been a paucity of effective exercise training studies in African American women; none have employed HIIT which appears uniquely suited given their metabolic profile and none have examined the impact of training on the metabolic response to an increase in dietary fat.

Therefore the Aims of this study are to determine, in overweight and obese, sedentary, pre-menopausal, non-diabetic African American women, whether a 14-week of a HIIT exercise program will:

I. Increase systemic post-absorptive lipid oxidation in response to a higher fat diet (50% fat, 35% CHO, 15% protein). The study team hypothesizes that the women who successfully complete training will have significantly higher post-absorptive lipid oxidation in response to the higher fat diet compared to the sedentary controls on a similar diet.

II. Improve aerobic endurance capacity. The study team hypothesizes that VO2peak will be significantly higher in the women who successfully complete training compared to the sedentary controls.

III. Improve insulin sensitivity. The study team hypothesizes that insulin sensitivity will be significantly higher in the women who successfully complete training compared to the sedentary controls.

Te secondary aims are to determine whether: 1) the exercise training favorably changes muscle adipose tissue distribution and lipid accumulation and 2) these changes correlate with an improvement in insulin sensitivity.

To test these hypotheses The study team will conduct a clinical trial in 48 pre-menopausal, healthy, sedentary, overweight and obese African American women. All women will be challenged with a 10-day eucaloric higher fat diet. Then, half of the women will be randomized to participate in a 14-week HIIT program designed to significantly increase their aerobic endurance and half will maintain baseline physical activity. Throughout the follow period all women will be counseled to follow the same, weight-maintaining, heart-healthy diet. After 14 weeks the higher fat dietary challenges will be repeated, at weight stability ensured with the use of the whole-body calorimeter (metabolic chamber). Post-absorptive lipid oxidation, insulin sensitivity and muscle-associated fat will be measured at the end of each of the higher fat diet periods, before and after the 14 weeks of exercise raining, in the sedentary and exercising women, 2 days after the last bout of acute exercise.

HIIT has a greater potential for translation into clinical practice as the shorter exercise time may improve compliance which is the biggest deterrent for the success of exercise training programs. Prevention of obesity and reversal of decreased aerobic capacity and insulin resistance in younger individuals such as African American women of child-bearing age (pre-menopausal) could be crucial to decrease the worrisome trends of obesity-related illnesses in African Americans.

ELIGIBILITY:
Inclusion Criteria:

* African American descent and all four grandparents reported as African Americans
* DNA will also be collected so admixture could be measured post study
* Reported good health (blood work, Hx and PE)
* Non-diabetic (OGTT)
* Pre-menopausal, Age range 20-40 years BMI range of 25-40, with regular menstrual periods
* Sedentary (exercise no more than 2 times/week, for one hour or spend no more than 1000 - 1500 Kcal/wk in physical activity as determined by a Paffenbarger questionnaire).

Exclusion Criteria:

* Any cardiac or pulmonary illnesses which may interfere with their capacity to exercise
* Active smoker
* Consume more than 2 oz. of ethanol/day
* Weight change greater than + 2 kg in the past 3 months
* Currently taking medications or have any physical conditions which may affect insulin action and/or lipid metabolism or have hyperlipidemia (plasma triglyceride greater than or equal to 350 mg/dl or total cholesterol levels greater than or equal to 300 mg/dl).
* Metal implants (ex: pacemaker, implanted jewelry, etc)
* 1st degree family history of type diabetes 2 diabetes (Will be noted but will not constitute an exclusionary criteria).

The subjects' usual diets will be evaluated by the Block 98.2 Food Frequency Questionnaire (BDDS, Berkeley, CA).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2013-04-16 (Actual); Study Completion 2013-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Post-absorptive Lipid Oxidation | Baseline and 14 weeks
  Resting ventilatory and gas exchange measurements will be done using indirect calorimetry using open circuit gas analysis at baseline and post intervention. Measurements and calculations for substrate utilization will be done as described and published using before and will be expressed as µmoles/KgFFM/min.

SECONDARY OUTCOMES:
Fitness (VO2peak) | up to 14 weeks
  All subjects will perform an incremental cycle ergometry test, at baseline and post intervention. The tests will be done before the 10-day eucaloric dietary challenges periods and data will be also used to determine the dietary prescription.
Glucose Disposal Rate (GDR) during the Hyperinsulinemic-Euglycemic Clamp | up to 14 weeks
  The subjects will be admitted at the CRR's inpatient physiology room to perform a Hyperinsulinemic-Euglycemic Clamp . The protocol used will be specific for measurements of insulin- mediated glucose disposal of the muscle. For 3 hours, plasma insulin concentration will be raised to around 200µU/ml using an insulin infusion of 80mU/m2 and the investigators will maintain euglycemia at around 100 mg/dl plasma glucose using a variable infusion of exogenous glucose of known concentration (20% glucose). Hepatic glucose production is expected to be completely suppressed at this level of insulin for these obese, but otherwise generally healthy women.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine Albu, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai St. Luke's Clinical Research Unit, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arad AD, Albu JB, DiMenna FJ. Feasibility of a progressive protocol of high-intensity interval training for overweight/obese, sedentary African American women: a retrospective analysis. BMC Sports Sci Med Rehabil. 2020 Sep 21;12:59. doi: 10.1186/s13102-020-00207-7. eCollection 2020. PMID 32974034